CLINICAL TRIAL: NCT03175874
Title: AVP Study: Autophagy and Pathological Aging Human Study in Osteoporosis With or Without Dementia of Alzheimer's Type
Brief Title: Autophagy and Pathological Aging
Acronym: AVP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-PP-03
Record Dates: First submitted 2017-05-29; First posted 2017-06-05 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Alzheimer Disease
MeSH Terms: conditions — Osteoporosis; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Quantification of autophagy (LC3II and SQSTM1 / p62) by Western blotting of purified OST proteins from a bone sample from resected femoral heads during laying of a total hip prosthesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- osteoporosis and alzheimer (Other): patient with osteoporosis and alzheimer hospitalized for total hip prosthesis.
  Interventions: Procedure: Hip bone sampling
- osteoporosis without alzheimer (Other): Patient with osteoporosis without alzheimer hospitalized for total hip prosthesis.
  Interventions: Procedure: Hip bone sampling
- Patient with arthrosis without alzheimer (Other): Patient with arthrosis without alzheimer hospitalized for total hip prosthesis.
  Interventions: Procedure: Hip bone sampling

INTERVENTIONS:
Procedure: Hip bone sampling — Quantification of autophagy (LC3II and SQSTM1 / p62) by Western blotting of purified OST proteins from a bone sample

SUMMARY:
Autophagy is recognized as a central mechanism for the regulation of aging. . Osteoporosis (OA) and Alzheimer's disease (AD) are two forms of pathological aging, sometimes entangled, including an over-risk of OP in AD and degradation of cognitive functions after OP fracture, but the link between These two pathologies remain poorly understood.

The aim of this prospective pilot study is to evaluate the level of autophagy of osteocytes (OST) in postmenopausal women with OP and to explore the hypothesis that the defect of autophagy is one of the physiopathological links of the OP During the MA

DETAILED DESCRIPTION:
Autophagy is a ubiquitous cellular mechanism that degrades and recycles toxic waste from cells. It is recognized as a central mechanism for the regulation of aging. Osteoporosis (OA) and Alzheimer's disease (AD) are two forms of pathological aging, sometimes entangled, including an over-risk of OP in AD and degradation of cognitive functions after OP fracture, but the link between These two pathologies remain poorly understood. In Alzheimer's disease (AD), a deficiency of autophagy is found both clinically and fundamentally. In animal studies, animal studies have shown that autophagy is involved in the differentiation, function and survival of bone cells, decreases with age and that a defect in autophagy is accompanied by a decrease in The bone mass. To date, we do not have human data on the autophagic capacities of bone cells in OP and AD.

The aim of this prospective pilot study is to evaluate the level of autophagy of osteocytes (OST) in postmenopausal women with OP and to investigate the hypothesis that the defect of autophagy is one of the physiopathological links of the OP During the MA.

The main objective is to determine, in two subgroups with or without Alzheimer's disease, whether there is an association between bone status and the level of autophagy of OST in postmenopausal women (OP versus non-OP)

Secondary objectives are to determine whether there is an association between the level of autophagy of the OST and the bone parameters (bone mineral density, serum vitamin D) and to compare in OP women the level of autophagy of the OST Of AM patients vs no MA.

Study population: Postmenopausal women over the age of 65 benefiting from the implantation of a hip prosthesis: 30 with an OP fracture of the femoral neck (15 non-MA and 15 MA, the cognitive status being determined by MMSE And IADL 1 month after the fracture) and 30 controls performed for osteoarthritis, free from OP (antecedents + bone mineral density) and MA (MMSE and IADL).

Primary endpoint: Quantification of autophagy (LC3II and SQSTM1 / p62) by Western blotting of purified OST proteins from a bone sample from resected femoral heads during laying of a total prosthesis Of hip.

Secondary endpoints: Bone mineral density of femoral neck and total hip (T-score and g / cm²) measured by X-ray biphotonic absorptiometry (Hologic QDR 4500) and serum 25 OH vitamin D (ng / ml).

Expected benefits: to better understand the role of autophagy in the pathophysiology of post-menopausal OP and AD in human pathology. Ultimately, it could potentially contribute to the design of new therapeutics targeting autophagy in the management of osteoporosis and more generally pathological aging.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for both groups:

* Women > 65 y: 2 groups

Inclusion criteria for Osteoporosis group (Alzheimer and non-Alzheimer):

* Osteoporotic femoral neck fracture requiring hip remplacement and fullfilling WHO definition of osteoporosis. Without any cognitive impairment for the first subgroup (MMSE > 26 and normal IADL) and with a final diagnosis of alzheimer disease in the other subgroup (DSM-IV-TR)

Inclusion criteria for Control group:

* Non osteoporotic (no fragility fracture (clinical or on VFA) and bone mineral density T-score > 2.5 SD at all sites)
* No cognitive impairment (MMSE > 26 and normal IADL)

Exclusion Criteria:

Non-Inclusion Criteria for both groups:

* Other pathologies associated with autophagy: Parkinson's disease, Crohn's disease, cancers, myopathies, type 2 diabetes
* Méd Medications interfering with autophagy: current corticosteroids, parathyroid hormone, estrogen, chloroquine, hydroxychloroquine, lithium, metformin, bisphosphonates,
* Dementia of non-Alzheimer type

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Quantification of autophagy | at inclusion
  Quantification of autophagy (LC3II and SQSTM1 / p62) by Western blotting of purified OST proteins from a bone sample from resected femoral heads

SECONDARY OUTCOMES:
Bone mineral density | at inclusion
  Bone mineral density of femoral neck and total hip (T-score and g / cm²) as measured by X-ray biphotonic absorptiometry (Hologic QDR 4500)
25 OH vitamin D (ng/ml). | at inclusion
  25 OH vitamin D (ng/ml) in serum

CONTACTS AND LOCATIONS:
Overall Officials: Veronique BREUIL, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- BREUIL, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Trojani MC, Clave A, Bereder I, Camuzard O, Bernard De Dompsure R, Gonzalez JF, Trojani C, Santucci-Darmanin S, Carle GF, Breuil V, Pierrefite-Carle V. Autophagy markers are decreased in bone of osteoporotic patients: a monocentric comparative study. Eur J Endocrinol. 2024 Mar 2;190(3):K27-K31. doi: 10.1093/ejendo/lvae017. PMID 38430550